CLINICAL TRIAL: NCT04639102
Title: Practical Alternative to Hospitalization
Acronym: PATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Independence Blue Cross (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 844436
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Emergency Department; Health, Subjective; Health Care Utilization
MeSH Terms: conditions — Emergencies; Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PATH Intervention (Experimental): Patients in the treatment arm will receive a personalized plan of care upon discharge from the emergency department.
  Interventions: Other: PATH Intervention
- Routine Care (No Intervention): Patients in the control arm will receive standard-of-care services (the care plan that the emergency physician would normally offer if PATH were not available) without PATH enrollment.

INTERVENTIONS:
Other: PATH Intervention — Patients will receive an enhanced level of care and service:
  1. Discharge planning- PATH clinicians will develop an individualized treatment plan at time of ED discharge. Each patient will receive next-day phone call to monitor status. There will be additional patient and family education, triage of new or worsening symptoms, and additional telephone contact as determined in treatment plan. There will be communication with home health teams as needed.
  2. Care coordination- PATH clinicians will arrange necessary primary medical doctor and specialty appointments. They will also communicate treatment plan to outpatient provider and arrange transportation for patients.
  3. Home monitoring/ Home Health Services- If patients are eligible and consent to home health services, they will be enrolled in Penn Medicine Home Health (PMHH). This will include virtual home monitoring, skilled nurse care, home physical and occupational therapists, social work services, and wound care.
  Arms: PATH Intervention

SUMMARY:
The investigators test the PATH program to evaluate whether the program allows patients to spend more days at home in comparison to patients who receive regular care. The program will involve patients from Penn Presbyterian Medical Center with a set of diagnoses and will provide patients with enhanced services upon discharge from the emergency department.

DETAILED DESCRIPTION:
The PATH program seeks to provide patients with enhanced services upon discharge from the emergency department, including visiting home nurses, visiting home physical and occupational therapists, scheduled frequent telephone visits with a medical provider, care coordination to arrange outpatient evaluation and testing, social work services, and other services. The purpose of this study is to evaluate whether the PATH program allows patients to spend more days at home in comparison to patients who receive regular care.

The broad goal of this program is to provide patients with a personalized package of enhanced services following discharge from the emergency department. In some cases, patients enrolled in the PATH program are likely to be discharged home regardless of enrollment, but are deemed potentially high-risk for returning to the hospital due to their illness or other factors. In other cases, enrolled patients might otherwise have been hospitalized but decide with their clinician that recovery at home is possible with the increased supervision and care provided by PATH. For all patients, we seek to determine whether PATH is effective in expediting patient recovery from acute illness and reduce the time spent in hospital or nursing facilities.

ELIGIBILITY:
Inclusion Criteria:

* Stable (Patients are deemed stable by ED clinician and PATH clinician per review of vital signs, history, exam, test results, and functional status)
* Have active insurance
* Domiciled at home (Patients must live in the community and not in nursing facility, shelter, or otherwise homeless)
* Safe home environment
* Live in Penn Medicine Home Health (PMHH) geographic catchment if enrolled in PMHH services

Exclusion Criteria:

* Substance use disorder (No active untreated SUD, including alcohol, opioids, cocaine, or stimulants)
* Serious mental health condition
* Police custody
* Homelessness
* Anticipated procedures or surgeries
* IV access (Patients with need for home infusion services or frequent blood testing after discharge must have standard level of IV access)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Days at home over 30 days | 30 days
  The number 30 minus the amount of days that patients spend in a hospital, nursing facility, or ED after discharge from the initial ED visit
Days that patients are expired | 30 days
  The number of days that patients are expired

SECONDARY OUTCOMES:
Impact of PATH on hospital operations - Capture rate | 5 months
  Percentage of eligible patients enrolled into the program (capture rate)
Quality of life at 30 days | 5 months
  This will be measured using the EQ-5D-5L questionnaire. This questionnaire measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each level is rated on scale that describes the degree of problems in that area.
Functional status at 30 days | 5 months
  This will be measured using the Lawton and Brody Instrumental Activities of Daily Living (Lawton-Brody IADL) Scale. This instrument assesses independent living skills and functional ability with 8 questions, including behaviors like telephoning, shopping, food preparation, housekeeping, laundering, use of transportation, use of medicine, and financial behavior.
  The scale is scored dichotomously (0= less able, 1= more able). The higher the score, the greater the person's abilities. Women are scored on all 8 areas of function, but, for men, the areas of food preparation, housekeeping, laundering are excluded. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women, and 0 to 5 for men.
Estimated cost (allowed charges) based on healthcare utilization | 5 months
  This will be determined by calculating allowed charges for healthcare services delivered to patient over 30-day follow up period.
Impact of PATH on hospital operations - percentage of hospitalized patients | 5 months
  Measured by potential eligible hospitalizations (patients screened as eligible if more likely to have been hospitalized from the ED); actual avoided hospitalizations (patients more likely to have been hospitalized from the ED who are enrolled in either treatment or control arm); and actual avoided hospitalizations (patients more likely to have been hospitalized from the ED and enrolled in the treatment arm).

CONTACTS AND LOCATIONS:
Overall Officials: Austin Kilaru, MD, MSHP, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No